CLINICAL TRIAL: NCT03762668
Title: Performance Assessment of a Modified Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLP691-C002
Record Dates: First submitted 2018-12-01; First posted 2018-12-04 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Refractive Errors; Myopia; Hyperopia
Keywords: Contact lens; Vision correction; Visual acuity
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MDACL, then DACL (Other): Modified delefilcon A contact lenses (MDACL) worn first, followed by delefilcon A contact lenses (DACL), as randomized. Each product worn bilaterally (in both eyes) for approximately 1 week in a daily disposable modality.
  Interventions: Device: Modified delefilcon A contact lenses; Device: Delefilcon A contact lenses
- DACL, then MDACL (Other): DACL worn first, followed by MDACL, as randomized. Each product worn bilaterally for approximately 1 week in a daily disposable modality.
  Interventions: Device: Modified delefilcon A contact lenses; Device: Delefilcon A contact lenses

INTERVENTIONS:
Device: Modified delefilcon A contact lenses — Spherical soft daily disposable contact lens
  Other Names: MDACL
Device: Delefilcon A contact lenses — Spherical soft daily disposable contact lens
  Other Names: DACL

SUMMARY:
The purpose of this study is to compare visual acuity between two daily disposable contact lenses.

DETAILED DESCRIPTION:
The expected duration of subject participation in the study is approximately 2 weeks, with 3 scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an approved Informed Consent form;
* Current wearer of commercial DAILIES TOTAL1 Contact Lenses in both eyes;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any eye condition that contraindicates contact lens wear, as determined by the Investigator;
* Any eye surgery that contraindicates contact lens wear, as determined by the Investigator;
* Wears habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week)
* Monocular (only one eye with functional vision);
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. CDMA Project Lead, Vision Care, Study Director — Alcon Research
Locations (5):
- United States (5):
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, West Palm Beach, Florida
  - Alcon Investigative Site, Ann Arbor, Michigan
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 investigative sites located in the United States.
Pre-assignment Details: Of the 62 subjects enrolled, 2 were exited as screen failures prior to randomization. This reporting group includes all randomized and exposed subjects (60).
Groups:
- MDACL, Then DACL: Modified delefilcon A contact lenses (MADCL) worn first, followed by delefilcon A contact lenses (DACL), as randomized. Each product worn bilaterally (in both eyes) for approximately 1 week in a daily disposable modality.
Period: Period 1, First Week of Wear
Arm/Group | MDACL, Then DACL | DACL, Then MDACL
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2, Second Week of Wear
Arm/Group | MDACL, Then DACL | DACL, Then MDACL
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects/eyes exposed to any study lens evaluated in this study (Safety Analysis Set).
Groups:
- MDACL, Then DACL: MDACL worn first, followed by DACL, as randomized. Each product worn bilaterally for approximately 1 week in a daily disposable modality.
- Total: Total of all reporting groups
Arm/Group | MDACL, Then DACL | DACL, Then MDACL | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.3) | 30.7 (8.6) | 31.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 29 | 26 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Distance Visual Acuity (logMAR)
Description: Distance visual acuity (VA) testing was performed using letter charts. Each row of the chart contained 5 letters, with the letters on each row progressively smaller than the row above. The subject read the letters from larger to smaller. The test terminated when the subject either misidentified a majority of letters on 1 row or progressed to the smallest row of letters. Visual acuity scoring sheets were used to record the number of letters correctly read. LogMAR VA was calculated based on the total number of letters read incorrectly as follows: LogMAR Acuity = base reading + (0.02 x number of letters missed). A lower logMAR value indicates better VA.
Time Frame: Day 1 Dispense, Day 7 Follow-Up
Population: All randomized subjects who were exposed to any study lenses evaluated in the study (Full Analysis Set), with non missing data.
Measure: Mean (Standard Deviation); unit: logMar
Units Other Than Participants: eyes
Groups:
- MDACL: MDACL worn for approximately 1 week, Period 1 or Period 2, as randomized
- DACL: DACL worn for approximately 1 week, Period 1 or Period 2, as randomized
Arm/Group | MDACL | DACL
Number analyzed (Participants) | 59 | 60
Number analyzed (eyes) | 118 | 120
logMar
  Day 1 Dispense | -0.04 (0.07) | -0.04 (0.07)
  Day 7 Follow-Up: number analyzed (Participants) | 59 | 59
  Day 7 Follow-Up: number analyzed (eyes) | 118 | 118
  Day 7 Follow-Up | -0.05 (0.07) | -0.05 (0.07)
Statistical Analysis 1: Comparison: MDACL vs DACL; Test type: Non-Inferiority — Noninferiority in VA was declared if the Upper Confidence Limit was less than 0.05; mixed effects repeated measures model; Least Squares Mean Difference = -0.00, 95% CI 1-sided [upper limit 0.01], Standard Error of Mean 0.005 — test minus control

ADVERSE EVENTS:
Time Frame: Adverse events were collected (observed or reported) for the duration of the individual's participation in the study, approximately 2 weeks.
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the study lenses. This analysis population includes all subjects/eyes exposed to any study lens evaluated in this study (Safety Analysis Set).
Arm/Group | MDACL | DACL
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT03762668/SAP_000.pdf
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT03762668/Prot_001.pdf